CLINICAL TRIAL: NCT01171430
Title: Assessment of Dynamic Contrast Enhanced Whole Body MRI (DCE-WB-MRI) as Independent Prognostic Factor for Disease-free Survival in Multiple Myeloma (After Intensification Therapy and Autologous Stem Cell Transplantation Suppressed by Amendment n°3)
Brief Title: "WB-DCE-MRI" in Multiple Myeloma as an Independent Prognostic Factor for Disease-free Survival
Acronym: EVALICEMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P081236
Record Dates: First submitted 2010-06-23; First posted 2010-07-28 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI WHOLE BODY (Experimental)
  Interventions: Device: Whole Body Dynamic Contrast Enhanced MRI (WB-DCE-MRI)

INTERVENTIONS:
Device: Whole Body Dynamic Contrast Enhanced MRI (WB-DCE-MRI) — 3 Whole Body Dynamic Contrast Enhanced MRI:
  * 1 WB-DCE-MRI before induction of chemotherapy(initial MRI).
  * 1 WB-DCE-MRI after induction high dose therapy and before intensification of chemotherapy and auto-transplant of hematopoietic sterns cells (early MRI).
  * 1 WB-DCE-MRI 3 months after treatment whatever (amendment n°3) (delayed MRI).
  Other Names: Mult.Myeloma eligible for Autologous Stem Cell Transpl.

SUMMARY:
The main objective of this study is to examine if absence of a satisfactory response on DCE-WB-MRI (see MR criteria of responders section) after completion of HDT followed by autologous stem-cell transplantation (ASCT) is an independent prognostic factor for EFS in patients with MM, compared with established ones including beta2-microglobulin and cytogenetic abnormalities. Secondary objectives are to examine if the microcirculation parameters obtained from baseline DCE-WB-MRI have prognostic significance and to examine if early DCE-WB-MRI performed after the induction HDT and before ASCT might also provide independent prognostic information for patient outcome, which might help in patient stratification and be integrated into the response criteria in the future.

DETAILED DESCRIPTION:
Introduction Bone marrow angiogenesis is increased in multiple myeloma (MM) and is an important prognostic factor for survival. Newly diagnosed MM patients have higher microvessel density (MVD) than controls on bone marrow biopsies. In addition, patients with higher MVD, receiving conventional chemotherapy or high-dose therapy with autologous stem cell transplantation, have shorter median overall survival than those with lower MVD by using the median MVD as the cutoff. In a study with 81 patients with MM treated with thalidomide with or without dexamethasone, MVD decreased significantly in responders while no significant change in MVD was seen in those failing to respond to thalidomide.

Microcirculation variables derived from dynamic contrast-enhanced magnetic resonance (DCE-MR) imaging, i.e. maximum enhancement and the exchange rate constant, correlate well with the histologic infiltration grade, MVD and serum markers of disease activity. Recently, the maximal amplitude of lumbar bone marrow enhancement on DCE-MR examination has been identified as a prognostic variable for event-free survival (EFS) in progressive MM. These parameters may serve as non-invasive surrogate biomarkers for determining prognosis and for assessing treatment response in myeloma patients. However, these studies used techniques which were limited to a maximal 400-mm field of view, whereas myeloma can involve the bone marrow focally, diffusely throughout the body, or even outside the marrow space. With the advancement of MR technologies, unenhanced whole-body MR imaging has proven more reliable than radiological skeletal survey and whole-body multidetector computed tomography in patients with MM.

Recently, whole-body single-phase contrast-enhanced sequence was applied in combination with unenhanced sequences for the detection of myeloma lesions. However, single-phase post-contrast MR examinations do not provide detailed enhancement curves, and this limitation possibly hinders the assessment of disease activity. On the other hand, segmental dynamic MR examinations do not enable assessment of the dynamic enhancement of focal lesions in different bone marrow segments. That was the reason which led us to develop a dynamic contrast-enhanced whole-body magnetic resonance imaging (DCE-WB-MRI) protocol, which was never explored in MM.

The treatment of patients with MM was largely palliative until, with the advent of high-dose melphalan, high rates of complete response (CR) could be obtained. For previously untreated patients aged 70 years (amendment n°5)or younger, high-dose therapy (HDT) followed by treatment (amendment n°3) with growth-factor-mobilized peripheral-blood stem cells (PBSCs) have been demonstrated superior to conventional chemotherapy with not only higher CR rates but also significantly extending EFS and overall survival. Recently, the International Myeloma Working Group proposed new uniform response criteria to facilitate precise comparisons between new evolving treatment strategies. As a functional imaging providing parameters related to angiogenesis and disease activity in MM, DCE-WB-MRI might provide additional information on prognostically important microcirculation variables on a whole-body scale. It might also prove helpful in assessing treatment response and further treatment strategy decision for patients with oligo- or nonsecretory disease.

Study Description :

Treatment regimen: the HDT followed by ASCT with PBSCs will be given. The ASCT will be conditioned by high-dose melphalan (HDMel) 200 mg/m2 with or without bortezomib following the actual guidelines.

Response assessment: clinical response will be assessed on the same day of each post-treatment MR examination and recorded according to the uniform response criteria. After completion of HDT followed by ASCT, patients will be followed every 4 months for the first two years and every 6 months thereafter for a total of at least 5 years. An event is defined as disease progression, relapse from clinical CR/VGPR, or death from any cause.

DCE-WB-MRI schedule: three MR examinations will be performed, the first at diagnosis and before initiation of chemotherapy, the second after induction chemotherapy and before ASCT, and the third exam three months after ASCT. The results of each DCE-WB-MRI will not influence further treatment strategy.

MR Criteria of Responders:

A satisfactory response on DCE-WB-MRI is defined by the presence of a maximal percentage of bone marrow enhancement below 100%. All focal lesions, if present, must not present an early enhancement but a progressive, delayed type maximal enhancement.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred to one of the hematology departement associated with the research project, with confirmed multiple myeloma defined according to uniform international criteria.
* Whatever stage classification according to Salmon and Durie with a life expectancy of more than 3 months.
* Age under 70 years old (amendment n°5) and eligible for autologous stem cell transplantation.
* Free and informed consent.

Exclusion Criteria:

* Patient unfit physically, mentally or legally to give informed consent.
* Patient non affiliate with social security scheme
* Patient with myeloma without measurable monoclonal immunoglobulin, including measurement of serum free light chains.
* Patient with another malignancy excluding basal cell cancer.
* Patient who could not undergo MRI (incompatible metallic foreign body, pacemaker, allergy to contrast, claustrophobia despite premedication, pregnancy, renal failure with creatinine clearance <30 ml/min

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Maximal percentage of bone marrow measurement on last WB DCE MRI | Measurements will be performed on initialWB DCE MRI Examination. Follow-up = Five year
  Bone marrow enhancement : Enhancement (%) = (SIpost - SIpre) x 100/SIpre, where SIpre is the signal intensity before injection and SIpost is the signal intensity after injection

SECONDARY OUTCOMES:
Maximal percentage of bone marrow measurement on initial WB DCE MRI | Measurements will be performed on initialWB DCE MRI Examination. Follow-up = Five year
  Bone marrow enhancement : Enhancement (%) = (SIpost - SIpre) x 100/SIpre, where SIpre is the signal intensity before injection and SIpost is the signal intensity after injection

CONTACTS AND LOCATIONS:
Overall Officials: Alain Luciani, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France